CLINICAL TRIAL: NCT01819051
Title: A Single Center, Pilot Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of the Plasma Treatment System in Treating Onychomycosis
Brief Title: Pilot Study to Evaluate Plasma Treatment of Onychomycosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moe Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOE - 131
Record Dates: First submitted 2013-03-22; First posted 2013-03-27 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

ARMS (1):
- Plasma (Experimental): Apply plasma to great toenail for up to 20 minutes, 1X/week for 3 weeks
  Interventions: Device: MOE Antimicrobial Plasma Treatment System

INTERVENTIONS:
Device: MOE Antimicrobial Plasma Treatment System — Plasma applied to great toenail 1X/week for three weeks

SUMMARY:
The purpose of this study is to evaluate the safety of treating human toenails with atmospheric plasma (MOE Antimicrobial Plasma Treatment System) and get an initial evaluation of the efficacy of this treatment for toenail fungus (onychomycosis).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 18 and 75 years of age inclusive, of either sex, and of any race;
* Subject must have distal subungual infection that affects approximately 25% to 50% of at least one great toenail, both clinically and mycologically diagnosed;
* Subject must have at least 2 mm of the proximal end of the target toenail free of infection;
* Subject must have a target toenail that is assessed as capable of growing approximately 1 mm/month, (e.g., the subject needs to report cutting his or her toenails at least once per month);
* Subject must be willing to give written informed consent and able to adhere to procedures and visit schedules;
* Woman of childbearing potential who is currently sexually active must agree to use a medically accepted method of contraception while receiving protocol-specified medication and for 30 days after stopping the medication. Methods include condoms (male or female) with or without a spermicidal agent, diaphragm or cervical cap with spermicide, medically prescribed intrauterine device, oral or systemic hormonal contraceptive (plus an additional reliable barrier method), and surgical sterilization (e.g., hysterectomy or tubal ligation).
* Woman of child-bearing potential who is not currently sexually active must agree to use a medically accepted method of contraception should she become sexually active while participating in the study.
* Woman of childbearing potential must have a negative serum pregnancy test within 72 hours prior to start of study drug.

Exclusion Criteria:

* Subject with one or more of the following conditions on the target toenail:
* proximal subungual onychomycosis,
* white superficial onychomycosis,
* dermatophytoma or "yellow spike/streak",
* exclusively lateral disease,
* inability to become normal in the opinion of the investigator.
* Subject with psoriasis, severe moccasin-type tinea pedis requiring treatment, symptomatic interdigital tinea pedis, lichen planus, or other abnormalities that could result in a clinically abnormal nail;
* Subject with peripheral vascular disease or peripheral circulatory impairment;
* Subject with history of uncontrolled diabetes mellitus;
* Subject with known chronic or active liver disease;
* Subject with any known immunodeficiency;
* Any pacemakers, or any metallic implants or prostheses in the vicinity of the treatment site (such as ankle, foot, etc.).
* Subject with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with study evaluations or optimal participation in the study;
* Subject who has received systemic antifungal therapy within 6 months or topical antifungal therapy applied to the foot or toenails within 1 month of study entry;
* Subject who has received radiation therapy, chemotherapy, and/or immunosuppressive drugs within 6 months of study, and/or oral corticosteroids for >1 month within the 6 months of study (exception: inhaled steroids);
* Subject known to have received treatment with investigational drugs within 30 days prior to enrollment into this study;
* Subject who is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function
* Subjects who may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse (no testing required), or subjects who are unable to return for scheduled follow-up visits
* Woman who is breastfeeding, pregnant, or intends to become pregnant;
* Subject who is part of the staff personnel directly involved with this study;
* Subject who is a family member of the investigational study staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in number of reported adverse events | Change from Baseline to 6 months post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College, New York, New York, United States